CLINICAL TRIAL: NCT03137823
Title: Diagnosis of GABHS Tonsillitis - Comparison Between Culture From Tonsills and Culture From the Bucal Surface
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bait Balev Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0022-17-BBL
Record Dates: First submitted 2017-03-16; First posted 2017-05-03 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Tonsillitis; Tonsillitis Streptococcal
Keywords: diagnosis, tonsillitis, streptococcus, GABHS
MeSH Terms: conditions — Tonsillitis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients (Other): each patient will be reviewed twice - first time culture from the tonsills and the second culture from the bucal surface.
  Interventions: Diagnostic Test: throat culture

INTERVENTIONS:
Diagnostic Test: throat culture — throat culture - from the tonsills and from the bucal surface

SUMMARY:
Diagnosis of Group A beta hemolytic strep tonsillitis -

* cultre of tonsills (gold standard)
* culture from bucal surface (test)

DETAILED DESCRIPTION:
This study will examine 2 groups. first group of 50 children aged 3-18 years and the second group of adults aged 18-65 with a clinical diagnosis of tonsillitis and centor criteria of 2 or more (fever, exudates on tonsills, no cough, enlarged lymph nodes).

In each patient we'll take 2 cultures - the first from the tonsills and the second from the bucal surface. both of them will be sent to MEGA-LAB .

the treatment will be based only on the gold standrad culture from the tonsills.

ELIGIBILITY:
Inclusion Criteria:

* tonsills exudates
* Centor criteria - 2 or more

Exclusion Criteria:

* tonsillectomy

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-05-22 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
positiveGABHS culture from bucal surface in comparisson to positive culture from tonsills | each test will be cultures within 24-48 hours.
  sensitivity and specificity of culture

CONTACTS AND LOCATIONS:
Locations (1):
- MACCABI, Ofakim, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adler L, Parizade M, Koren G, Yehoshua I. Oral cavity swabbing for diagnosis of group a Streptococcus: a prospective study. BMC Fam Pract. 2020 Mar 26;21(1):57. doi: 10.1186/s12875-020-01129-6. PMID 32216750